CLINICAL TRIAL: NCT01346852
Title: Predictive Ability of Therapeutic Risk Factors in Pediatric and Adult Asthma Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112607
Record Dates: First submitted 2011-04-15; First posted 2011-05-03 (Estimated); Results first posted 2011-06-01 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: pediatrics; Medicaid; asthma; outcomes; asthma medication ratio
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pediatric participants: Pediatric participants (age 4 to 17) with a diagnosis of asthma
  Interventions: Drug: Asthma treatment with an asthma-related medication and at least one asthma controller medication
- Adult participants: Adult participants (age 18 and older) with a diagnosis of asthma
  Interventions: Drug: Asthma treatment with an asthma-related medication and at least one asthma controller medication

INTERVENTIONS:
Drug: Asthma treatment with an asthma-related medication and at least one asthma controller medication — participants with an asthma diagnosis who also had at least one dispensing event of an asthma-related medication and had at least one asthma controller medication (inhaled corticosteroids containing inhalers, methylxanthines, leukotriene receptor antagonists, cromolyn sodium) or albuterol.

SUMMARY:
The purpose of this study is to assess the predictive ability of three asthma risk markers: the ratio of controller medication to total asthma medication, an albuterol only marker, and an oral corticosteroid use marker, as well as to compare the precision of these tools between adult and pediatric patient populations. This retrospective longitudinal analysis will use 2 different databases: a large managed care database and a large fee for service Medicaid database.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with asthma as determined by ICD-9 codes and asthma drug use
* at least 4 years of age
* use of at least 1 controller or at least 5 albuterol prescriptions in 12 months

Exclusion Criteria:

* Subjects with COPD or treatment for COPD

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study intends to identify subjects at least 4 years of age with asthma and using asthma medications
Sampling Method: Probability Sample
Enrollment: 101437 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric Participants Diagnosed With Asthma: Pediatric (4-17 years old) participants with an asthma diagnosis who also had at least one dispensing event of an asthma-related medication during the enrollment period (January 1, 2004 to June 30, 2006) and had at least one asthma controller medication (inhaled corticosteroids containing inhalers, methylxanthines, leukotriene receptor antagonists, cromolyn sodium) or albuterol. Due to the retrospective nature of this analysis, doses received and frequency of dosing are not known.
- Adult Participants Diagnosed With Asthma: Adult (>=18 years old) participants with an asthma diagnosis who also had at least one dispensing event of an asthma-related medication during the enrollment period (January 1, 2004 to June 30, 2006) and had at least one asthma controller medication (inhaled corticosteroids containing inhalers, methylxanthines, leukotriene receptor antagonists, cromolyn sodium) or albuterol. Due to the retrospective nature of this analysis, doses received and frequency of dosing are not known.
Period: Overall Study
Arm/Group | Pediatric Participants Diagnosed With Asthma | Adult Participants Diagnosed With Asthma
Started | 41753 | 59684
Completed | 41753 | 59684
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Participants Diagnosed With Asthma | Adult Participants Diagnosed With Asthma | Total
Number analyzed (Participants) | 41753 | 59684 | 101437
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.1 (4.0) | 43.6 (13.3) | 29.8 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18339 | 38211 | 56550
  Male | 23414 | 21473 | 44887

OUTCOME MEASURES:

1. Primary Outcome: Mean Ratio of Controller Medication to Total Asthma Medication
Description: The ratio of controller medication (CM) to total asthma medication (AM), which is well established in predicting future asthma events in adults, was calculated as the ratio of the units of CMs used during the defined period divided by the sum of the units of CMs plus the units of inhaled short-acting beta-agonists used during the same period. A CM is defined as any inhaled corticosteroid containing medication, methylxanthines, leukotriene receptor antagonists, or cromolyn sodium. The ratio is calculated using all CM. Asthma controllers are medications used to treat asthma on a regular basis.
Time Frame: January 1, 2004 to June 30, 2006: 3, 6, and 12 month follow-up periods
Population: Ingenix Impact National Managed Care Database members who had >=1 ICD-9 code for asthma and had >= 1 controller medication or >=5 albuterol canisters dispensed identified in the database during the 12-month identification period (pre-index). We tested 3 different capture/follow-up periods; thus, sample sizes varied depending capture period used.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pediatric Participants Diagnosed With Asthma | Adult Participants Diagnosed With Asthma
Number analyzed (Participants) | 40659 | 59174
ratio
  3 months, n=40419, 59016 | 0.57 (0.34) | 0.66 (0.34)
  6 months, n=40525, 59091 | 0.66 (0.26) | 0.71 (0.29)
  12 months, n=40659, 59174 | 0.63 (0.26) | 0.70 (0.29)

2. Secondary Outcome: Mean Number of Short-acting Beta-agonist (SABA) Canisters Used
Description: The number of albuterol canisters dispensed is a marker that is well established in predicting future asthma events in an adult population.
Time Frame: January 1, 2004 to June 30, 2006: 3, 6, and 12 month follow-up periods
Population: Ingenix Impact National Managed Care Database members who had >=1 ICD-9 code for asthma and had >= 1 controller medication or >=1 albuterol canister dispensed during the 12-month pre-index period.
Measure: Mean (Standard Deviation); unit: canisters
Arm/Group | Pediatric Participants Diagnosed With Asthma | Adult Participants Diagnosed With Asthma
Number analyzed (Participants) | 41753 | 59684
canisters
  3 months | 1.03 (0.90) | 1.04 (1.06)
  6 months | 1.24 (1.18) | 1.28 (1.57)
  12 months | 1.72 (1.86) | 1.82 (2.71)

ADVERSE EVENTS:
Description: This was a retrospective observational study using a large health insurance claims database. Serious adverse events and non-serious adverse events were not collected.
Arm/Group | Pediatric Participants Diagnosed With Asthma | Adult Participants Diagnosed With Asthma
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.